CLINICAL TRIAL: NCT02729350
Title: The Feasibility of the PAINReportIt Guided Relaxation Intervention for Pain and Stress in Adult Inpatients With Sickle Cell Disease
Brief Title: The Feasibility of the PAINReportIt Guided Relaxation Intervention-INPATIENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201500671
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease; Stress; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Relaxation video clip (Experimental): This intervention is a 12-minute guided audio-visual relaxation intervention delivered at the baseline (Day 1) visit to determine the immediate effects of guided relaxation intervention on stress and pain in inpatients with sickle cell disease. The GR intervention also includes six video clips, ranging from 2 to 20 minutes in length to determine the short-term (Day 5) effects of guided relaxation intervention on stress and pain.
  Interventions: Behavioral: Guided Relaxation video clip
- Sickle cell experience discussion (Other): Attention Control Group: This intervention is a 12-minute sickle cell disease experience discussion. In this computer-based discussion, patients will discuss their experience of having sickle cell disease. The audio-taped questions and onscreen directions were programmed to be self-administered. Subjects' responses will be captured via the microphone so that Data Collectors are not involved in this discussion process, and it is equivalent to the guided relaxation activity.
  Interventions: Behavioral: Sickle Cell Disease Experience Discussion

INTERVENTIONS:
Behavioral: Guided Relaxation video clip — This intervention is a 12-minute guided relaxation intervention for reducing pain and stress in adult inpatients with sickle cell disease.
  Arms: Guided Relaxation video clip
Behavioral: Sickle Cell Disease Experience Discussion — This intervention is a 12-minute sickle cell disease experience discussion.
  Arms: Sickle cell experience discussion

SUMMARY:
The goal of this research study is to improve the self-management of pain, stress, and cognitive/affective symptoms that may result in adult inpatients with sickle cell disease (SCD) by determining the feasibility of a self-management guided relaxation (GR) stress reduction intervention using a tablet-based mobile device. Currently, opioid analgesics are primarily used to treat SCD pain while self-managed behavioral modalities such as GR, are rarely used, particularly, in inpatient settings. Little is known about the effects or mechanisms of GR on pain, stress, and cognitive/affective symptoms in adults with SCD hospitalized with pain. Emerging evidence from the hypothalamic pituitary adrenal (HPA) axis theory offer insights for understanding the mechanisms. Adding GR as a supplement to analgesic therapies will address the dearth of self-management strategies for controlling pain in SCD. GR is a simple and cost-effective non-drug intervention that could reduce pain and stress in inpatients with SCD. GR is an intervention where inpatients with SCD are directed to listen to and view audio-visual recordings while they visualize themselves being immersed in that scenario.

DETAILED DESCRIPTION:
The purpose of this research study is to see if a new computerized stress reduction program, called PAINReportIt Guided Relaxation Intervention, can be used to teach people who have sickle cell disease (SCD) how to track their stress and pain daily and use guided audio-visual relaxation exercises to help them reduce their stress and pain. To obtain preliminary data for a larger trial, 30 adult inpatients with SCD admitted with SCD pain will be recruited.

The investigators will stratify patients on worst pain intensity (<=5 and >5) and randomly assign 15 adults to Attention Control (12-min SCD experience discussion on Day 1 and daily stress/pain tracking on Days 2-4) and 15 adults to Experimental (12-min GR video clip on Day 1 and daily stress/pain tracking and GR on Days 2-4) groups.

Immediate effects on pain, stress, and relaxation responses after the 12-min session will be examined. Patients will continue the trial for additional 4 days, with self-management on Days 2-4 and posttest on Day 5 while hospitalized to test short-term effects.

During Days 2-4, the experimental group will choose and watch any of six video clips (2 min, 5 min, 8 min, 10 min, 15 min, and 20 min lengths) at least once a day; and at stress onset and as often as they need. We will investigate mechanisms by which GR produces its effects in adult inpatients with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Has SCD diagnosis;
* Reports pain 3 or greater in the previous 24 hours (0-10 scale)
* admitted to University of Florida (UF) Health for pain crisis
* Speaks and reads English
* 18 years of age or older
* self-identifies as being of African descent or Hispanic

Exclusion Criteria:

* Legally blind
* Physically or cognitively unable to complete study measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Current Pain | Immediate (Day 1 baseline) and Day 2-5
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain intensity scale: A 3-item scale that asks patients to report their pain now, worst, and average on a scale of 1 to 5 where 1 is "had no pain" and 5 is "very severe." We will estimate intervention effects using regression analysis.
Average pain intensity | Short-term (Day 5)
  PAINReportIt® Pain intensity scale: A 3-item scale that asks patients to report their current, least, and worst pain intensity today, on a scale of 0 to 10, where 0 is "no pain" and 10 is "pain as bad as it could be." We will average the three scores to create an average pain intensity score. We will estimate intervention effects using linear regression.
Composite pain index | Short-term (Day 5)
  PAINReportIt® Composite pain index (CPI): A a multidimensional representation of pain calculated by averaging the individual proportional scores for each of the four pain dimensions: (1) number of pain sites; (2) pain intensity; (3) total pain rating index (from the McGill Pain Questionnaire [MPQ], pain quality); and (4) pain pattern score. The scores for the CPI range from 0 to 100. We will estimate intervention effects using linear regression.

SECONDARY OUTCOMES:
Current stress | Immediate (Day 1 baseline) and Days 2-5
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We will estimate intervention effects using linear regression.
Average stress intensity | Short-term (Day 5)
  Stress intensity scale: A 3-item scale that asks patients to report their current, least, and worst stress intensity today, on a scale of 0 to 10, where 0 is "no stress" and 10 is "stress as bad as it could be." We will average the three scores to create an average stress intensity score. We will estimate intervention effects using linear regression.

OTHER OUTCOMES:
Physiologic markers of relaxation (pulse, respiration, finger temperature) | Immediate (baseline)
  Physiological markers of relaxation (pulse, respiration, finger temperature) will be measured using a standard vital sign measuring device. We expect to observe trends for the immediate GR effect in terms of decreases in relaxation indicators (respiration rate, heart rate) and increases in skin temperature. We will estimate intervention effects using regression analysis.
Level of relaxation | Immediate (Day 1 baseline) and Day 2-5
  Relaxation rating scale. A 1-item scale that asks patients to report their level of relaxation on a scale of 0 to 10, where 0 is "not at all relaxed" and 10 is "completely relaxed." We will estimate intervention effects using linear regression.
Perceived stress | Baseline
  Perceived Stress Questionnaire: A 30-item questionnaire that measures perceived stress in the last two weeks. An overall perceived stress index (PSI) score for each scale is computed by subtracting 30 from the raw score and dividing it by 90, yielding scores that range from 0 to 1. Higher scores indicate greater perceived stress recent. We will analyze data using linear regression.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam O Ezenwa, PhD, RN, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No